CLINICAL TRIAL: NCT06880302
Title: Male Infertility and Assisted Reproductive Technologies Research Biobank
Acronym: MARK
Status: Recruiting | Type: Observational
Sponsor: Reproductive Medicine Associates of New Jersey (Other)
Responsible Party: Sponsor
Other Study IDs: RMA-2022-01
Record Dates: First submitted 2025-03-11; First posted 2025-03-17 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Male Infertility; Infertility (IVF Patients)
MeSH Terms: conditions — Infertility, Male; Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Specimens include testicular tissue, sperm, semen samples, donor sperm or discarded sperm preps. Buccal swabs will also be collected if participants decide to participate in sub-study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Males providing specimen for infertility treatment: Males providing specimen for infertility treatment

SUMMARY:
The objective of this research is to build a biobank of biological male specimens used for diagnostics and treatment of infertility or assisted reproductive technologies (ART).

DETAILED DESCRIPTION:
The objective of this research is to build a biobank of biological male specimens used for diagnostics and treatment of infertility or assisted reproductive technologies (ART). These specimens include testicular tissue, sperm, semen samples, donor sperm or discarded sperm preps. These samples were possibly utilized for diagnostic testing such as semen analyses or DNA fragmentation testing or for ART procedures such as intrauterine insemination (IUI) in-vitro fertilization (IVF) or intracytoplasmic sperm injection (ICSI) and are no longer needed clinically. Rather than discarding those samples the men who provided them or the sperm recipient in the case of donor sperm may elect to donate them for future research purposes. These samples will be used for future research regarding male infertility and assisted reproductive technologies.

ELIGIBILITY:
Inclusion Criteria:

* Males providing testicular tissue, sperm, semen samples, discarded sperm preps for IUI/IVF/ICSI or the sperm recipient for those utilizing donor sperm, for cryopreservation at the respective site(s) for either clinical use or preservation

Exclusion Criteria:

* Samples that are quarantined or in isolation dewars for infectious diseases

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Males that had previously provided male biological specimen for their infertility treatment that no longer wishes to keep their samples frozen
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-03-04 (Actual); Primary Completion 2032-04 (Estimated); Study Completion 2032-12 (Estimated)

PRIMARY OUTCOMES:
Biobank | 5 years
  The purpose of this study is to create a biobank of male biological specimens

CONTACTS AND LOCATIONS:
Locations (1):
- RMANJ, Basking Ridge, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No